CLINICAL TRIAL: NCT02135692
Title: A Multi-Centre, Open-Label, Study of Mepolizumab in a Subset of Subjects With a History of Life Threatening/Seriously Debilitating Asthma Who Participated in the MEA115661 Trial
Brief Title: A Phase 3a, Repeat Dose, Open-label, Long-term Safety Study of Mepolizumab in Asthmatic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201312; 2014-000314-54 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Asthma
Keywords: Severe eosinophilic asthma; Extension study; Expanded access; Safety; Mepolizumab; Eosinophils
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mepolizumab 100 mg (Experimental): All subjects will receive mepolizumab 100mg administered SC into the upper arm or thigh approximately every 4 weeks.
  Interventions: Biological: Mepolizumab; Drug: SOC

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab is a fully humanised IgG antibody (IgG1, kappa) with human heavy and light chain frameworks. Mepolizumab will be supplied as a lyophilised cake in sterile vials for individual use.
Drug: SOC — Standard of Care (SOC) will differ by participant, however it will generally include oral corticosteroids and an inhaled controller medicine (an inhaled corticosteroid plus a long acting beta agonist) and/or short acting beta agonists

SUMMARY:
This is a multi-center, open-label, long-term study of subcutaneously (SC) administered mepolizumab 100mg in addition to standard of care (SOC), in subjects with severe eosinophilic asthma. This study will enroll a subset of subjects from Study MEA115661 who have demonstrated clear benefit from therapy and who without continuation of mepolizumab therapy are individuals at greatest risk of serious deterioration of their health status. In order to target individuals at greatest risk for serious deterioration of their health status, only subjects from the MEA115661 study with a history of life-threatening or seriously debilitating asthma, will be allowed to participate. Subjects meeting all of the eligibility criteria for the study will be offered the opportunity to consent for this study of up to 128 weeks in length (including the Follow-Up Visit). This study will give opportunity to extend the collection of clinical data for long-term use and further assess the sustainability of efficacy in a population likely to experience significant loss of asthma control and the need for higher doses of systemic steroids if returned to SOC only.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Prior to commencing any study related activities, subjects must be able and willing to provide written informed consent.
* Male or Eligible Female Subjects: To be eligible for the study, females of child-bearing potential must commit to consistent and correct use of an acceptable method of birth control and for 4 months after the last study drug administration. A urine pregnancy test is required of all females of childbearing potential at the initial Baseline Visit (Visit 1).
* French Subjects Only: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.
* MEA115661 Participation: Subjects must have completed Visit 14 of MEA115661.
* Current Anti-Asthma Therapy: The subject's asthma has been treated with an ICS controller medication for the last 8 months with fluticasone propionate (FP) >=500 mcg/day (or equivalent).
* Disease Severity: Subjects must be assessed as having life-threatening /serious debilitating asthma in order to enroll, as defined by the following: Subjects enrolled in MEA115588 must meet one of the following criteria: a) Subject has a history of at least one intubation during their lifetime; b) >=3 asthma exacerbations in the 12 months prior to screening for MEA115588; c) >=1 or more hospitalization for asthma exacerbation in the 12 months prior to screening for MEA115588. Subjects enrolled in MEA115575 must meet one of the following criteria: d) Subject has a history of at least one intubation during their lifetime; e) Their optimized dose at randomization in MEA115575 was >=10mg of prednisone; f) >=1 or more hospitalization for asthma exacerbation in the 12 months prior to screening for MEA115575.
* Clinical Benefit: Subjects must have experienced documented clinical benefit to enroll. Subjects must meet the following criteria demonstrating clinical benefit: Subjects enrolled in MEA115588 who received mepolizumab must meet all of the following criteria: a) Subject must have had a reduction in their exacerbation frequency by >=50% during MEA115588. The baseline for comparison is the total number of exacerbations reported in the 12 months prior to screening for MEA115588. b) The investigator response on the "Clinician-Rated Response to Therapy" questionnaire at Visit 10 was either: mildly improved, moderately improved or significantly improved. Subjects enrolled in MEA115588 who received placebo must meet all of the following criteria: c) Subject must have had a reduction in their exacerbation frequency by >=50% during the first 8 months of MEA115661. The baseline for comparison is the total number of exacerbations reported in the 12 months prior to screening for MEA115588; d) The investigator confirms that the subject demonstrated improvement during MEA115661. Subjects enrolled in MEA115575 who received mepolizumab must meet all of the following criteria: e) Subject must have reduced their oral corticosteroid dose by >=50% during MEA115575. The baseline for comparison is the subject's optimized oral corticosteroid (OCS) dose at randomization in MEA115575; f) The investigator response on the "Clinician-Rated Response to Therapy" questionnaire at Visit 9 was either: mildly improved, moderately improved or significantly improved. Subjects enrolled in MEA115575 who received placebo must meet all of the following criteria: g) Subject must have reduced their oral corticosteroid dose at randomization by >=50% in the first 6 months of MEA115661. The baseline for comparison is the subject's optimized OCS dose at randomization in MEA115575; h) The investigator confirms that the subject demonstrated improvement during MEA115661.

Exclusion Criteria

* Health Status: Clinically significant change in health status during MEA115661 which in the opinion of the investigator would make the subject unsuitable for participation in this long-term study.
* Pregnancy: Subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnanDeart during the time of study participation.
* Exacerbation History: Subjects who received placebo in MEA115588 and had NO exacerbations during the study.
* Oral Corticosteroid Use: Subjects who received placebo in MEA115575 and were able to discontinue oral corticosteroid therapy by the end of the study.
* Smoking Status: Current smokers
* Previous Significant Protocol Deviation: Subjects who were excluded from the per protocol analysis due to significant protocol deviations in either study MEA115575 or MEA115588.
* Electrocardiogram (ECG) Assessment: A clinically significant ECG abnormality at the exit visit of MEA115661, as determined by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (103):
- United States (16):
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Salt Lake City, Utah
- Argentina (5):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (4):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St-Charles-Borromée, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- Chile (3):
  - GSK Investigational Site, Rancagua, Reg Del Libert Bern Ohiggins
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Talcahuano
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- France (10):
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Strasbourg
- Germany (11):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Italy (7):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Pietra Ligure (SV), Liguria
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Cittadella PD, Veneto
- Japan (9):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leeuwarden
- Poland (2):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
- Russia (3):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Korea (6):
  - GSK Investigational Site, Anyang-Si Gyeonggi-do
  - GSK Investigational Site, Bucheon City, Gyenggi-do
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Donggu Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
- Spain (3):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
- Ukraine (4):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Vinnytsia
- United Kingdom (4):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20059

REFERENCES:
- [Background] Khurana S, Brusselle GG, Bel EH, FitzGerald JM, Masoli M, Korn S, Kato M, Albers FC, Bradford ES, Gilson MJ, Price RG, Humbert M. Long-term Safety and Clinical Benefit of Mepolizumab in Patients With the Most Severe Eosinophilic Asthma: The COSMEX Study. Clin Ther. 2019 Oct;41(10):2041-2056.e5. doi: 10.1016/j.clinthera.2019.07.007. Epub 2019 Aug 22. PMID 31447130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, long-term study of mepolizumab 100 milligram (mg) administered subcutaneously (SC), in addition to standard of care (SOC), in eligible participants with severe eosinophilic asthma, who completed the MEA115661 Exit Visit (Visit 14). The study enrolled participants across 18 countries.
Pre-assignment Details: A total of 340 participants were screened for the study, of which one participant was screening failure, and 339 participants received the study treatment.
Groups:
- Mepolizumab 100 mg SC: Participants received mepolizumab 100 mg administered via SC injection into the upper arm or thigh approximately every 4 weeks for 172 weeks. Participants remained on standard of care asthma therapy which could be adjusted during the study at the discretion of the physician.
Period: Overall Study
Arm/Group | Mepolizumab 100 mg SC
Started | 339
Completed | 0
Not Completed | 339
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 2
Not completed — Subject met Liver Stopping Criteria | 1
Not completed — Product commercially available | 159
Not completed — Study closed/terminated | 153
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ Ethnicity: Asian-Central/South Asian Heritage | 2
  Race/ Ethnicity: Asian-East Asian Heritage | 19
  Race/ Ethnicity: Asian-Japanese Heritage | 26
  Race/ Ethnicity: Asian-South East Asian Heritage | 4
  Race/ Ethnicity: Black or African American | 4
  Race/ Ethnicity: White-Arabic/North African Heritage | 7
  Race/ Ethnicity: White-White/Caucasian/European Heritage | 277

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of On-treatment Exacerbations Per Year
Description: Exacerbations are defined as the worsening of asthma which requires use of systemic corticosteroids intravenous (IV) or oral steroid like prednisone, for at least 3 days or a single intramuscular (IM) corticosteroid (CS) dose is required. For maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visit. On-Treatment data between first dose date and earliest of Withdrawal date/last dose + 28 days was considered for analysis. Analysis of the number of exacerbations was performed using a negative binomial generalized linear model.
Time Frame: Baseline (Week 0) to Week 172
Population: As Treated (AT) Population. AT Population included all participants who received at least one dose of mepolizumab within study 201312.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Exacerbations per year | 0.93 [0.81 to 1.06]

2. Primary Outcome: Number of Participants With Any On-treatment Adverse Event (AE) or On-treatment Serious AE (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. On-treatment AEs and on-treatment SAEs are the events occurring on/after the first dose of open-label mepolizumab date and before/on last dose+28 days.
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Participants
  Any AE | 315
  Any SAE | 84

3. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire (ACQ)-5 On-treatment Score
Description: The ACQ-5 is a five-item questionnaire developed as a measure of participants asthma control. The five questions enquire about the frequency and/or severity of symptoms (nocturnal awakening on waking in the morning, activity limitation, shortness of breath, wheeze). The response options for all these questions consist of a 0 (no impairment/limitation) to 6 (total impairment/ limitation) scale. The overall ACQ score is calculated as the mean of the 5 questions and therefore ranges between 0 (totally controlled) and 6 (severely uncontrolled). Baseline was considered as the latest assessment prior to first dose of mepolizumab in this study. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value.
Time Frame: Baseline (Week 0) to Week 168
Population: AT Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Scores on a scale
  Week 12, n=333: number analyzed (Participants) | 333
  Week 12, n=333 | -0.16 (1.096)
  Week 24, n=333: number analyzed (Participants) | 333
  Week 24, n=333 | -0.15 (1.131)
  Week 36, n=326: number analyzed (Participants) | 326
  Week 36, n=326 | -0.21 (1.089)
  Week 48, n=328: number analyzed (Participants) | 328
  Week 48, n=328 | -0.17 (0.965)
  Week 60, n=307: number analyzed (Participants) | 307
  Week 60, n=307 | -0.18 (1.066)
  Week 72, n=282: number analyzed (Participants) | 282
  Week 72, n=282 | -0.08 (1.145)
  Week 84, n=254: number analyzed (Participants) | 254
  Week 84, n=254 | -0.03 (1.151)
  Week 96, n=212: number analyzed (Participants) | 212
  Week 96, n=212 | -0.12 (0.976)
  Week 108, n=190: number analyzed (Participants) | 190
  Week 108, n=190 | -0.06 (1.057)
  Week 120, n=164: number analyzed (Participants) | 164
  Week 120, n=164 | -0.01 (1.244)
  Week 132, n=135: number analyzed (Participants) | 135
  Week 132, n=135 | -0.09 (1.089)
  Week 144, n=73: number analyzed (Participants) | 73
  Week 144, n=73 | 0.34 (1.220)
  Week 156, n=23: number analyzed (Participants) | 23
  Week 156, n=23 | 0.07 (0.962)
  Week 168, n=6: number analyzed (Participants) | 6
  Week 168, n=6 | -0.33 (0.935)

4. Secondary Outcome: Mean Change From Baseline in On-treatment Clinic Pre-bronchodilator FEV1
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry at Baseline and Weeks 24, 48, 72, 96, 120, 144 and 168. Spirometry was performed within 1 hour of the Baseline assessment. Baseline was considered as the latest assessment prior to first dose of mepolizumab in this study. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). Data between first dose date and earliest of Withdrawal date/last dose + 28 days considered on-treatment.
Time Frame: Baseline (Week 0) to Week 168
Population: AT Population
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Milliliter
  Week 24, n=332: number analyzed (Participants) | 332
  Week 24, n=332 | 67 (382.9)
  Week 48, n=325: number analyzed (Participants) | 325
  Week 48, n=325 | 27 (404.6)
  Week 72, n=289: number analyzed (Participants) | 289
  Week 72, n=289 | 30 (406.0)
  Week 96, n=223: number analyzed (Participants) | 223
  Week 96, n=223 | 47 (433.7)
  Week 120, n=169: number analyzed (Participants) | 169
  Week 120, n=169 | 34 (369.9)
  Week 144, n=88: number analyzed (Participants) | 88
  Week 144, n=88 | 14 (374.9)
  Week 168, n=15: number analyzed (Participants) | 15
  Week 168, n=15 | 78 (302.9)

5. Secondary Outcome: Number of Participants Withdrawn From the Study Due to Lack of Efficacy and Adverse Events
Description: AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Number of participants withdrawn due to lack of efficacy and adverse events from the study have been presented.
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Participants
  Withdrawals due to lack of efficacy | 2
  Withdrawals due to adverse events | 3

6. Secondary Outcome: Number of Participants Hospitalized Due to Adverse Events Including Asthma Exacerbations
Description: AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia. Number of participants requiring hospitalization due to an on-treatment serious adverse event including asthma exacerbations are presented. On-treatment SAEs are the events occurring on/after the first dose of mepolizumab date and before/on last dose of mepolizumab + 28 days.
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Participants | 78

7. Secondary Outcome: Number of Participants With AEs Including Both Systemic (Allergic and Non-allergic) and Local Site Reactions
Description: AEs were collected from the Baseline visit until the follow-up visit (Week 172). Participants were monitored to evaluate the AEs of systemic and local site reaction. AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. On treatment AEs were defined as events occurring from the first dose until 28 days after the last dose of mepolizumab. Number of participants with AEs including both systemic (i.e. allergic/immunoglobulin (Ig)E-mediated and non-allergic) and local site reactions have been presented.
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Participants
  Any systemic events | 2
  Any local site reactions | 14

8. Secondary Outcome: Mean Change From Baseline in QT Interval Corrected by Bazett's Method (QTcB) and QT Interval Corrected by Fridericia's Method (QTcF) Values for 12-lead Electrocardiogram (ECG)
Description: Twelve-lead ECG measurements were recorded after the participant has rested in the supine position for 5 minutes. The ECG was obtained before lung function testing followed by other study procedures. Baseline was considered as the latest assessment prior to first dose of mepolizumab in this study. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles)..
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Milliseconds
  QTcB, Week 24, n=301: number analyzed (Participants) | 301
  QTcB, Week 24, n=301 | 0.1 (16.90)
  QTcB, Week 48, n=294: number analyzed (Participants) | 294
  QTcB, Week 48, n=294 | -0.9 (17.27)
  QTcB, Week 72, n=269: number analyzed (Participants) | 269
  QTcB, Week 72, n=269 | -2.9 (18.13)
  QTcB, Week 96, n=221: number analyzed (Participants) | 221
  QTcB, Week 96, n=221 | -0.6 (17.96)
  QTcB, Week 144, n=131: number analyzed (Participants) | 131
  QTcB, Week 144, n=131 | 0.5 (21.07)
  QTcB, Week 172, n=16: number analyzed (Participants) | 16
  QTcB, Week 172, n=16 | 1.8 (22.08)
  QTcF, Week 24, n=301: number analyzed (Participants) | 301
  QTcF, Week 24, n=301 | -1.1 (14.61)
  QTcF, Week 48, n=294: number analyzed (Participants) | 294
  QTcF, Week 48, n=294 | -1.3 (14.08)
  QTcF, Week 72, n=269: number analyzed (Participants) | 269
  QTcF, Week 72, n=269 | -3.7 (15.68)
  QTcF, Week 96, n=221: number analyzed (Participants) | 221
  QTcF, Week 96, n=221 | -0.8 (16.18)
  QTcF, Week 144, n=131: number analyzed (Participants) | 131
  QTcF, Week 144, n=131 | -0.0 (17.88)
  QTcF, Week 172, n=16: number analyzed (Participants) | 16
  QTcF, Week 172, n=16 | 1.7 (17.06)

9. Secondary Outcome: Number of Participants With Maximum Change From Baseline in QTcB and QTcF Interval for ECG Assessed at Any Time Post Baseline
Description: Twelve-lead ECG measurements were recorded after the participant has rested in the supine position for 5 minutes. The ECG was obtained before lung function testing followed by other study procedures. Baseline was considered as the latest assessment prior to first dose of mepolizumab in this study. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value. Participants with maximum change from Baseline were summarised at any time post Baseline for the following categories <-60, >=-60 to <-30, >=-30 to <0, >=0 to <30, >=30 to <60 and >=60. QTc intervals shown at any time post Baseline are the maximum seen in each participant over the course of the trial.
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 305
Participants
  QTcB, <-60 | 0
  QTcB, >=-60 to <-30 | 1
  QTcB, >=-30 to < 0 | 70
  QTcB, >= 0 to < 30 | 196
  QTcB, >= 30 to < 60 | 35
  QTcB, >=60 | 3
  QTcF, <-60 | 0
  QTcF, >=-60 to <-30 | 1
  QTcF, >=-30 to < 0 | 77
  QTcF, >= 0 to < 30 | 199
  QTcF, >= 30 to < 60 | 28
  QTcF, >=60 | 0

10. Secondary Outcome: Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure
Description: Vital sign measurements including systolic blood pressure (SBP) and diastolic blood pressure (DBP) were done pre-injection with the participants sitting, having rested in this position for at least 5 minutes before each reading. They were taken before measurement of any clinic lung function tests or ECGs at the specified time point. Baseline was considered as the latest assessment prior to first dose of mepolizumab in this study. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value.
Time Frame: Baseline (Week 0) to Week 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Millimeter of mercury
  SBP, Week 4, n=333: number analyzed (Participants) | 333
  SBP, Week 4, n=333 | 1.8 (11.26)
  SBP, Week 8, n=334: number analyzed (Participants) | 334
  SBP, Week 8, n=334 | 0.6 (11.75)
  SBP, Week 12, n=337: number analyzed (Participants) | 337
  SBP, Week 12, n=337 | 1.5 (12.48)
  SBP, Week 16, n=334: number analyzed (Participants) | 334
  SBP, Week 16, n=334 | 2.0 (12.35)
  SBP, Week 20, n=327: number analyzed (Participants) | 327
  SBP, Week 20, n=327 | 1.2 (13.69)
  SBP, Week 24, n=333: number analyzed (Participants) | 333
  SBP, Week 24, n=333 | 1.8 (13.35)
  SBP, Week 28, n=330: number analyzed (Participants) | 330
  SBP, Week 28, n=330 | 1.4 (13.56)
  SBP, Week 32, n=324: number analyzed (Participants) | 324
  SBP, Week 32, n=324 | 1.0 (13.43)
  SBP, Week 36, n=330: number analyzed (Participants) | 330
  SBP, Week 36, n=330 | 0.8 (13.00)
  SBP, Week 40, n=327: number analyzed (Participants) | 327
  SBP, Week 40, n=327 | 1.6 (13.44)
  SBP, Week 44, n=327: number analyzed (Participants) | 327
  SBP, Week 44, n=327 | 1.2 (12.75)
  SBP, Week 48, n=329: number analyzed (Participants) | 329
  SBP, Week 48, n=329 | 1.8 (13.22)
  SBP, Week 52, n=325: number analyzed (Participants) | 325
  SBP, Week 52, n=325 | 1.5 (13.31)
  SBP, Week 56, n=324: number analyzed (Participants) | 324
  SBP, Week 56, n=324 | 2.0 (13.52)
  SBP, Week 60, n=315: number analyzed (Participants) | 315
  SBP, Week 60, n=315 | 2.0 (13.17)
  SBP, Week 64, n=307: number analyzed (Participants) | 307
  SBP, Week 64, n=307 | 2.5 (13.37)
  SBP, Week 68, n=286: number analyzed (Participants) | 286
  SBP, Week 68, n=286 | 2.5 (13.46)
  SBP, Week 72, n=281: number analyzed (Participants) | 281
  SBP, Week 72, n=281 | 2.3 (13.35)
  SBP, Week 76, n=274: number analyzed (Participants) | 274
  SBP, Week 76, n=274 | 2.3 (12.31)
  SBP, Week 80, n=265: number analyzed (Participants) | 265
  SBP, Week 80, n=265 | 3.5 (13.58)
  SBP, Week 84, n=255: number analyzed (Participants) | 255
  SBP, Week 84, n=255 | 2.7 (14.01)
  SBP, Week 88, n=245: number analyzed (Participants) | 245
  SBP, Week 88, n=245 | 1.5 (13.70)
  SBP, Week 92, n=218: number analyzed (Participants) | 218
  SBP, Week 92, n=218 | 0.7 (13.24)
  SBP, Week 96, n=208: number analyzed (Participants) | 208
  SBP, Week 96, n=208 | 1.2 (13.39)
  SBP, Week 100, n=199: number analyzed (Participants) | 199
  SBP, Week 100, n=199 | 1.0 (12.43)
  SBP, Week 104, n=197: number analyzed (Participants) | 197
  SBP, Week 104, n=197 | 2.4 (13.38)
  SBP, Week 108, n=192: number analyzed (Participants) | 192
  SBP, Week 108, n=192 | 1.7 (12.76)
  SBP, Week 112, n=182: number analyzed (Participants) | 182
  SBP, Week 112, n=182 | 1.8 (14.12)
  SBP, Week 116, n=177: number analyzed (Participants) | 177
  SBP, Week 116, n=177 | 1.9 (14.66)
  SBP, Week 120, n=167: number analyzed (Participants) | 167
  SBP, Week 120, n=167 | 1.9 (13.63)
  SBP, Week 124, n=152: number analyzed (Participants) | 152
  SBP, Week 124, n=152 | 2.5 (14.88)
  SBP, Week 128, n=151: number analyzed (Participants) | 151
  SBP, Week 128, n=151 | 2.6 (14.15)
  SBP, Week 132, n=139: number analyzed (Participants) | 139
  SBP, Week 132, n=139 | 1.0 (14.37)
  SBP, Week 136, n=112: number analyzed (Participants) | 112
  SBP, Week 136, n=112 | 2.3 (14.94)
  SBP, Week 140, n=91: number analyzed (Participants) | 91
  SBP, Week 140, n=91 | -0.9 (16.53)
  SBP, Week 144, n=77: number analyzed (Participants) | 77
  SBP, Week 144, n=77 | 2.3 (14.13)
  SBP, Week 148, n=62: number analyzed (Participants) | 62
  SBP, Week 148, n=62 | 0.6 (13.02)
  SBP, Week 152, n=35: number analyzed (Participants) | 35
  SBP, Week 152, n=35 | 0.6 (11.33)
  SBP, Week 156, n=32: number analyzed (Participants) | 32
  SBP, Week 156, n=32 | 1.5 (15.73)
  SBP, Week 160, n=14: number analyzed (Participants) | 14
  SBP, Week 160, n=14 | 4.4 (9.48)
  SBP, Week 164, n=8: number analyzed (Participants) | 8
  SBP, Week 164, n=8 | 7.0 (15.07)
  SBP, Week 168, n=1: number analyzed (Participants) | 1
  SBP, Week 168, n=1 | -4.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  DBP, Week 4, n=333: number analyzed (Participants) | 333
  DBP, Week 4, n=333 | 0.1 (8.41)
  DBP, Week 8, n=334: number analyzed (Participants) | 334
  DBP, Week 8, n=334 | -0.8 (8.81)
  DBP, Week 12, n=337: number analyzed (Participants) | 337
  DBP, Week 12, n=337 | 0.2 (9.25)
  DBP, Week 16, n=334: number analyzed (Participants) | 334
  DBP, Week 16, n=334 | 0.5 (9.30)
  DBP, Week 20, n=327: number analyzed (Participants) | 327
  DBP, Week 20, n=327 | -0.7 (10.35)
  DBP, Week 24, n=333: number analyzed (Participants) | 333
  DBP, Week 24, n=333 | -0.2 (9.40)
  DBP, Week 28, n=330: number analyzed (Participants) | 330
  DBP, Week 28, n=330 | 0.1 (8.88)
  DBP, Week 32, n=324: number analyzed (Participants) | 324
  DBP, Week 32, n=324 | -0.1 (10.44)
  DBP, Week 36, n=330: number analyzed (Participants) | 330
  DBP, Week 36, n=330 | -0.4 (10.12)
  DBP, Week 40, n=327: number analyzed (Participants) | 327
  DBP, Week 40, n=327 | -0.6 (9.24)
  DBP, Week 44, n=327: number analyzed (Participants) | 327
  DBP, Week 44, n=327 | 0.1 (9.39)
  DBP, Week 48, n=329: number analyzed (Participants) | 329
  DBP, Week 48, n=329 | 0.2 (9.71)
  DBP, Week 52, n=325: number analyzed (Participants) | 325
  DBP, Week 52, n=325 | -0.1 (9.83)
  DBP, Week 56, n=324: number analyzed (Participants) | 324
  DBP, Week 56, n=324 | 0.7 (9.77)
  DBP, Week 60, n=315: number analyzed (Participants) | 315
  DBP, Week 60, n=315 | -0.5 (10.40)
  DBP, Week 64, n=307: number analyzed (Participants) | 307
  DBP, Week 64, n=307 | -0.4 (9.92)
  DBP, Week 68, n=286: number analyzed (Participants) | 286
  DBP, Week 68, n=286 | -0.1 (10.04)
  DBP, Week 72, n=281: number analyzed (Participants) | 281
  DBP, Week 72, n=281 | -0.3 (10.13)
  DBP, Week 76, n=274: number analyzed (Participants) | 274
  DBP, Week 76, n=274 | -0.2 (9.92)
  DBP, Week 80, n=265: number analyzed (Participants) | 265
  DBP, Week 80, n=265 | 0.7 (9.83)
  DBP, Week 84, n=255: number analyzed (Participants) | 255
  DBP, Week 84, n=255 | -0.6 (10.05)
  DBP, Week 88, n=245: number analyzed (Participants) | 245
  DBP, Week 88, n=245 | -0.3 (9.22)
  DBP, Week 92, n=218: number analyzed (Participants) | 218
  DBP, Week 92, n=218 | -0.9 (9.10)
  DBP, Week 96, n=208: number analyzed (Participants) | 208
  DBP, Week 96, n=208 | -0.2 (9.17)
  DBP, Week 100, n=199: number analyzed (Participants) | 199
  DBP, Week 100, n=199 | -0.7 (10.04)
  DBP, Week 104, n=197: number analyzed (Participants) | 197
  DBP, Week 104, n=197 | 0.1 (10.21)
  DBP, Week 108, n=192: number analyzed (Participants) | 192
  DBP, Week 108, n=192 | 0.1 (9.89)
  DBP, Week 112, n=182: number analyzed (Participants) | 182
  DBP, Week 112, n=182 | 0.0 (10.17)
  DBP, Week 116, n=177: number analyzed (Participants) | 177
  DBP, Week 116, n=177 | -0.1 (10.31)
  DBP, Week 120, n=167: number analyzed (Participants) | 167
  DBP, Week 120, n=167 | 0.4 (9.74)
  DBP, Week 124, n=152: number analyzed (Participants) | 152
  DBP, Week 124, n=152 | -0.3 (11.11)
  DBP, Week 128, n=151: number analyzed (Participants) | 151
  DBP, Week 128, n=151 | 0.6 (9.58)
  DBP, Week 132, n=139: number analyzed (Participants) | 139
  DBP, Week 132, n=139 | -0.5 (10.10)
  DBP, Week 136, n=112: number analyzed (Participants) | 112
  DBP, Week 136, n=112 | 0.1 (9.89)
  DBP, Week 140, n=91: number analyzed (Participants) | 91
  DBP, Week 140, n=91 | -1.8 (9.68)
  DBP, Week 144, n=77: number analyzed (Participants) | 77
  DBP, Week 144, n=77 | -0.6 (10.92)
  DBP, Week 148, n=62: number analyzed (Participants) | 62
  DBP, Week 148, n=62 | -0.7 (11.03)
  DBP, Week 152, n=35: number analyzed (Participants) | 35
  DBP, Week 152, n=35 | -1.0 (8.97)
  DBP, Week 156, n=32: number analyzed (Participants) | 32
  DBP, Week 156, n=32 | -2.0 (10.42)
  DBP, Week 160, n=14: number analyzed (Participants) | 14
  DBP, Week 160, n=14 | 2.9 (7.92)
  DBP, Week 164, n=8: number analyzed (Participants) | 8
  DBP, Week 164, n=8 | 1.9 (8.06)
  DBP, Week 168, n=1: number analyzed (Participants) | 1
  DBP, Week 168, n=1 | 5.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.

11. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Vital sign measurements including pulse rate was done pre-injection with the participants sitting, having rested in this position for at least 5 minutes before each reading. They were taken before measurement of any clinic lung function tests or ECGs at the specified time point. Baseline was considered as the latest assessment prior to first dose of mepolizumab in this study. The change from Baseline is defined as the difference between the value of the endpoint at the time point of interest and Baseline value.
Time Frame: Baseline (Week 0) to Week 168
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Beats per minute
  Pulse rate, Week 4, n=334: number analyzed (Participants) | 334
  Pulse rate, Week 4, n=334 | 2.1 (9.98)
  Pulse rate, Week 8, n=333: number analyzed (Participants) | 333
  Pulse rate, Week 8, n=333 | 2.3 (10.65)
  Pulse rate, Week 12, n=337: number analyzed (Participants) | 337
  Pulse rate, Week 12, n=337 | 2.6 (11.05)
  Pulse rate, Week 16, n=334: number analyzed (Participants) | 334
  Pulse rate, Week 16, n=334 | 2.1 (11.03)
  Pulse rate, Week 20, n=327: number analyzed (Participants) | 327
  Pulse rate, Week 20, n=327 | 2.7 (11.10)
  Pulse rate, Week 24, n=333: number analyzed (Participants) | 333
  Pulse rate, Week 24, n=333 | 1.2 (11.22)
  Pulse rate, Week 28, n=330: number analyzed (Participants) | 330
  Pulse rate, Week 28, n=330 | 2.8 (10.43)
  Pulse rate, Week 32, n=324: number analyzed (Participants) | 324
  Pulse rate, Week 32, n=324 | 2.7 (11.44)
  Pulse rate, Week 36, n=330: number analyzed (Participants) | 330
  Pulse rate, Week 36, n=330 | 2.6 (11.02)
  Pulse rate, Week 40, n=327: number analyzed (Participants) | 327
  Pulse rate, Week 40, n=327 | 2.7 (11.09)
  Pulse rate, Week 44, n=327: number analyzed (Participants) | 327
  Pulse rate, Week 44, n=327 | 2.7 (12.05)
  Pulse rate, Week 48, n=329: number analyzed (Participants) | 329
  Pulse rate, Week 48, n=329 | 0.4 (10.63)
  Pulse rate, Week 52, n=325: number analyzed (Participants) | 325
  Pulse rate, Week 52, n=325 | 1.7 (10.48)
  Pulse rate, Week 56, n=324: number analyzed (Participants) | 324
  Pulse rate, Week 56, n=324 | 2.1 (11.36)
  Pulse rate, Week 60, n=315: number analyzed (Participants) | 315
  Pulse rate, Week 60, n=315 | 2.1 (10.97)
  Pulse rate, Week 64, n=307: number analyzed (Participants) | 307
  Pulse rate, Week 64, n=307 | 2.7 (10.96)
  Pulse rate, Week 68, n=286: number analyzed (Participants) | 286
  Pulse rate, Week 68, n=286 | 2.9 (11.32)
  Pulse rate, Week 72, n=281: number analyzed (Participants) | 281
  Pulse rate, Week 72, n=281 | 2.0 (11.15)
  Pulse rate, Week 76, n=274: number analyzed (Participants) | 274
  Pulse rate, Week 76, n=274 | 2.8 (11.15)
  Pulse rate, Week 80, n=265: number analyzed (Participants) | 265
  Pulse rate, Week 80, n=265 | 3.3 (11.45)
  Pulse rate, Week 84, n=255: number analyzed (Participants) | 255
  Pulse rate, Week 84, n=255 | 3.2 (12.21)
  Pulse rate, Week 88, n=245: number analyzed (Participants) | 245
  Pulse rate, Week 88, n=245 | 2.4 (11.98)
  Pulse rate, Week 92, n=218: number analyzed (Participants) | 218
  Pulse rate, Week 92, n=218 | 2.4 (12.42)
  Pulse rate, Week 96, n=208: number analyzed (Participants) | 208
  Pulse rate, Week 96, n=208 | 0.0 (11.16)
  Pulse rate, Week 100, n=199: number analyzed (Participants) | 199
  Pulse rate, Week 100, n=199 | 1.8 (12.30)
  Pulse rate, Week 104, n=197: number analyzed (Participants) | 197
  Pulse rate, Week 104, n=197 | 2.3 (12.29)
  Pulse rate, Week 108, n=192: number analyzed (Participants) | 192
  Pulse rate, Week 108, n=192 | 2.2 (11.34)
  Pulse rate, Week 112, n=182: number analyzed (Participants) | 182
  Pulse rate, Week 112, n=182 | 2.3 (12.35)
  Pulse rate, Week 116, n=177: number analyzed (Participants) | 177
  Pulse rate, Week 116, n=177 | 2.0 (12.06)
  Pulse rate, Week 120, n=167: number analyzed (Participants) | 167
  Pulse rate, Week 120, n=167 | 1.2 (12.19)
  Pulse rate, Week 124, n=152: number analyzed (Participants) | 152
  Pulse rate, Week 124, n=152 | 2.3 (12.56)
  Pulse rate, Week 128, n=151: number analyzed (Participants) | 151
  Pulse rate, Week 128, n=151 | 1.5 (11.69)
  Pulse rate, Week 132, n=139: number analyzed (Participants) | 139
  Pulse rate, Week 132, n=139 | 2.2 (12.46)
  Pulse rate, Week 136, n=112: number analyzed (Participants) | 112
  Pulse rate, Week 136, n=112 | 2.0 (11.68)
  Pulse rate, Week 140, n=92: number analyzed (Participants) | 92
  Pulse rate, Week 140, n=92 | 0.7 (11.45)
  Pulse rate, Week 144, n=77: number analyzed (Participants) | 77
  Pulse rate, Week 144, n=77 | -1.5 (11.92)
  Pulse rate, Week 148, n=62: number analyzed (Participants) | 62
  Pulse rate, Week 148, n=62 | -0.5 (11.68)
  Pulse rate, Week 152, n=35: number analyzed (Participants) | 35
  Pulse rate, Week 152, n=35 | -0.6 (13.80)
  Pulse rate, Week 156, n=32: number analyzed (Participants) | 32
  Pulse rate, Week 156, n=32 | -0.4 (12.94)
  Pulse rate, Week 160, n=14: number analyzed (Participants) | 14
  Pulse rate, Week 160, n=14 | 1.5 (13.24)
  Pulse rate, Week 164, n=8: number analyzed (Participants) | 8
  Pulse rate, Week 164, n=8 | 1.4 (21.23)
  Pulse rate, Week 168, n=1: number analyzed (Participants) | 1
  Pulse rate, Week 168, n=1 | 36.0 (NA) — NA indicates that data were not available as n=1 at this timepoint

12. Secondary Outcome: Number of Participants With Positive Anti-mepolizumab Binding Antibodies (ADA) and Neutralizing Antibodies (NAb)
Description: Blood samples were collected for the determination of ADA just prior to administration of mepolizumab. Samples that tested positive for anti-mepolizumab antibodies were further tested for the presence of NAb. The highest value post-Baseline visit are based on each participant's highest post-Baseline titer. NAb assay result was only presented for participants with positive ADA assay. Highest value post-Baseline would be positive for a participant who had both negative and positive post-Baseline results. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Participants
  Highest value post-Baseline, ADA, positive, n=335: number analyzed (Participants) | 335
  Highest value post-Baseline, ADA, positive, n=335 | 6
  Highest value post-Baseline, ADA, Negative, n=335: number analyzed (Participants) | 335
  Highest value post-Baseline, ADA, Negative, n=335 | 329
  Highest value post-Baseline, NAb, positive, n=6: number analyzed (Participants) | 6
  Highest value post-Baseline, NAb, positive, n=6 | 0
  Highest value post-Baseline, NAb, Negative, n=6: number analyzed (Participants) | 6
  Highest value post-Baseline, NAb, Negative, n=6 | 6

13. Secondary Outcome: Number of Participants With Potential Clinical Importance Values for Change From Baseline Relative to the Reference Range for Clinical Chemistry Parameters at Any Time Post-Baseline
Description: Blood samples were collected to assess clinical chemistry laboratory parameters. Number of participants with Potential Clinical Importance values for change from Baseline relative to the reference range at any time post-Baseline are presented. Any time post Baseline = all visits (including scheduled and unscheduled) post-Baseline. Participants are counted in the category that their value changes to (low, normal or high), unless there was no change in their category. If lab value category was unchanged, participants were recorded in the "To Normal or No Change" category. Alanine Aminotransferase=ALT. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 339
Participants
  Glucose, To low, n=336: number analyzed (Participants) | 336
  Glucose, To low, n=336 | 1
  Glucose, To Normal or No Change, n=336: number analyzed (Participants) | 336
  Glucose, To Normal or No Change, n=336 | 334
  Glucose, To high, n=336: number analyzed (Participants) | 336
  Glucose, To high, n=336 | 1
  ALT, To low, n=337: number analyzed (Participants) | 337
  ALT, To low, n=337 | 0
  ALT, To Normal or No Change, n=337: number analyzed (Participants) | 337
  ALT, To Normal or No Change, n=337 | 337
  ALT, To high, n=337: number analyzed (Participants) | 337
  ALT, To high, n=337 | 0
  Calcium, To low, n=336: number analyzed (Participants) | 336
  Calcium, To low, n=336 | 0
  Calcium, To Normal or No Change, n=336: number analyzed (Participants) | 336
  Calcium, To Normal or No Change, n=336 | 336
  Calcium, To high, n=336: number analyzed (Participants) | 336
  Calcium, To high, n=336 | 0
  Phosphate, To low, n=336: number analyzed (Participants) | 336
  Phosphate, To low, n=336 | 0
  Phosphate, To Normal or No Change, n=336: number analyzed (Participants) | 336
  Phosphate, To Normal or No Change, n=336 | 336
  Phosphate, To high, n=336: number analyzed (Participants) | 336
  Phosphate, To high, n=336 | 0
  Potassium, To low, n=336: number analyzed (Participants) | 336
  Potassium, To low, n=336 | 0
  Potassium, To Normal or No Change, n=336: number analyzed (Participants) | 336
  Potassium, To Normal or No Change, n=336 | 336
  Potassium, To high, n=336: number analyzed (Participants) | 336
  Potassium, To high, n=336 | 0
  Sodium, To low, n=336: number analyzed (Participants) | 336
  Sodium, To low, n=336 | 1
  Sodium, To Normal or No Change, n=336: number analyzed (Participants) | 336
  Sodium, To Normal or No Change, n=336 | 335
  Sodium, To high, n=336: number analyzed (Participants) | 336
  Sodium, To high, n=336 | 0

14. Secondary Outcome: Number of Participants With Potential Clinical Importance Values for Change From Baseline Relative to the Reference Range for Hematology Parameters at Any Time Post-Baseline
Description: Blood samples were collected to assess hematology laboratory parameters. Number of participants with Potential Clinical Importance values for change from Baseline relative to the reference range at any time post-Baseline are presented. Any time post Baseline = all visits (including scheduled and unscheduled) post-Baseline. Participants are counted in the category that their value changes to (low, normal or high), unless there was no change in their category. If lab value category was unchanged, participants were recorded in the "To Normal or No Change" category.
Time Frame: Baseline (Week 0) to Week 172
Population: AT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 336
Participants
  Hematocrit, To low | 1
  Hematocrit, To Normal or No Change | 335
  Hematocrit, To high | 0
  Hemoglobin, To low | 1
  Hemoglobin, To Normal or No Change | 335
  Hemoglobin, To high | 0
  Leukocytes, To low | 1
  Leukocytes, To Normal or No Change | 335
  Leukocytes, To high | 0
  Platelets, To low | 1
  Platelets, To Normal or No Change | 335
  Platelets, To high | 0

ADVERSE EVENTS:
Time Frame: The on-treatment AEs and on-treatment SAEs are the events which happened on/after the first dose of mepolizumab date and before/on last dose of mepolizumab date + 28 days (up to 172 weeks)
Description: AEs and SAEs were collected for all participants within the As Treated Population which comprised of all participants who received at least one dose of mepolizumab.
Arm/Group | Mepolizumab 100 mg SC
All-Cause Mortality (participants affected / at risk) | 2/339
Serious Adverse Events (participants affected / at risk) | 84/339
Other Adverse Events (participants affected / at risk) | 288/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 100 mg SC (N=339)
Asthma (Respiratory, thoracic and mediastinal disorders) | 34 (51)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (5)
Diverticulitis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Congenital anomaly (Congenital, familial and genetic disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 100 mg SC (N=339)
Nasopharyngitis (Infections and infestations) | 143 (270)
Bronchitis (Infections and infestations) | 64 (106)
Upper respiratory tract infection (Infections and infestations) | 64 (110)
Sinusitis (Infections and infestations) | 62 (115)
Influenza (Infections and infestations) | 42 (52)
Respiratory tract infection (Infections and infestations) | 20 (23)
Gastroenteritis (Infections and infestations) | 19 (20)
Lower respiratory tract infection (Infections and infestations) | 18 (28)
Rhinitis (Infections and infestations) | 18 (31)
Urinary tract infection (Infections and infestations) | 17 (19)
Pharyngitis (Infections and infestations) | 15 (22)
Ear infection (Infections and infestations) | 12 (15)
Viral upper respiratory tract infection (Infections and infestations) | 12 (14)
Pneumonia (Infections and infestations) | 11 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 52 (78)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (27)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (51)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (48)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (16)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Headache (Nervous system disorders) | 57 (160)
Dizziness (Nervous system disorders) | 15 (19)
Diarrhoea (Gastrointestinal disorders) | 16 (17)
Nausea (Gastrointestinal disorders) | 15 (16)
Vomiting (Gastrointestinal disorders) | 14 (32)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (13)
Fatigue (General disorders) | 16 (23)
Influenza like illness (General disorders) | 15 (17)
Injection site reaction (General disorders) | 15 (48)
Eczema (Skin and subcutaneous tissue disorders) | 14 (17)
Rash (Skin and subcutaneous tissue disorders) | 14 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (17)
Insomnia (Psychiatric disorders) | 17 (18)
Hypertension (Vascular disorders) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT02135692/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT02135692/SAP_001.pdf